CLINICAL TRIAL: NCT04856540
Title: Clinical Characteristic and Quality of Life Assessment in Adulthood of Patients With Cryopyrin Associated Periodic Syndrome
Brief Title: Adult Outcomes of Children With CAPS
Acronym: CAPS
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/0105; 2021-A00585-36 (Other: ID-RCB number,ANSM)
Record Dates: First submitted 2021-04-13; First posted 2021-04-23 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Cryopyrin Associated Periodic Syndrome
Keywords: CAPS Cryopyrin associated periodic syndromes; MWS Muckle-Wells syndrome; CINCA Chronic infantile neurological cutaneous and articular syndrome ;; FCAS Familial cold auto-inflammatory syndrome; Phenotype ; Quality of life; Quality of life
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The patients included in this study were followed up in the Internal Medicine and Paediatrics Departments of the Lille CHU, the Paediatric Rheumatology and Immunology Department of the Necker Enfant Malade Hospital in Paris and the Paediatric Rheumatology Department and Internal Medicine of the Bicêtre Hospital in Paris. All patients selected presented one of the 3 CAPS clinical phenotypes (CINCA/NOMID, Muckle-Wells or Cold Urticaria). The mutation and the determination of the variant had to be confirmed by genetic analysis.

Patient data were collected from their medical records, retrospectively. Data collected concern childhood period from appearance of symptoms, adulthood period, in the last year and patients' way of life and quality of life upon the assessment. In addition, we collected demographic data related to the patients' lifestyle (intoxications, living arrangements, level of education) and we conducted individual telephone interviews lasting 15 minutes to complete a quality of life questionnaire including the SF36 questionnaire.

The study aimed to describe the clinical symptoms of patients in adulthood and to assess quality of life. We also wanted to compare the clinical phenotypes of patients according to their genetic variant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FCAS, Muckle-Wells or NOMID/CINCA;
* age < 16 years at the apparition of the first symptoms of the disease;
* age ≥ 16 years old at inclusion
* follow-up in a CEREMAIA reference or competence center.

Exclusion Criteria:

* Age < 16 years at inclusion;
* non-consenting patient

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients follow-up in a CEREMAIA reference or competence center.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-02-25 (Actual); Study Completion 2022-02-25 (Actual)

PRIMARY OUTCOMES:
Clinical characteristics of patients with CAPS in adulthood | Baseline

SECONDARY OUTCOMES:
Assessment of the quality of life of patients with CAPS in adulthood | Baseline
Compare the clinical status between childhood and adulthood | Baseline
Compare the clinical status of patients according to their genetic variant. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hachulla, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- Hop Claude Huriez Chu Lille, Lille, France